CLINICAL TRIAL: NCT04117971
Title: Knowledge, Attitude and Practice of Child Abuse Diagnosis and Reporting Among a Group of Egyptian Dentists: A Cross Sectional Study
Brief Title: Knowledge, Attitude and Practice of Child Abuse Diagnosis and Reporting Among a Group of Egyptian Dentists
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nora Magdy Mahmoud Elsayed, Master's candidate, Cairo University
Other Study IDs: 14422017451433
Record Dates: First submitted 2019-10-04; First posted 2019-10-07 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Child Abuse
Keywords: Child abuse; Abuse diagnosis; Abuse report; dentists' knowledge
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Staff members: Staff members in different clinical departments at Faculty of Dentistry, Cairo University.
  Interventions: Other: Questionnaire
- PhD students: PhD candidates in different clinical departments at Faculty of Dentistry, Cairo University.
  Interventions: Other: Questionnaire
- Master's students: Master's candidates in in different clinical departments at Faculty of Dentistry, Cairo University.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — The study will involve structured questionnaire asking questions about knowledge, attitude, and practice of child abuse diagnosis and reporting among dentists.

SUMMARY:
Child abuse is defined as "Any act of commission or omission that endangers or impairs child's physical, sexual, or emotional health and development". According to The Centres for Disease Control and Prevention (CDC), Child physical abuse CPA is defined as "The intentional use of physical force against a child that result in, or has the potential to result in, physical injury".

Child abuse and neglect may occur in any family, and it isn't confined to certain geographic, ethnic, or socioeconomic background. According to World Health Organization (WHO) estimation, around forty million children suffer from different forms of abuse, and require health and social care.

WHO has estimated that in year 2000 nearly fifty-seven thousand children under fifteen years old were dead because of abuse, with the highest rate in children between zero to four years old. In 2014, WHO estimated that 23% of children worldwide were subjected to physical abuse.

Dentists are the best to detect children who are at abuse risk, since more than fifty percent of abuse injuries occur at head and neck region, and they are the first to see and treat orofacial region. Studies have shown that while dentists are in a good position to detect and report abuse, few of them do report abuse cases.

The main causes of not reporting CPA are lack of adequate history, inability, and hesitancy in diagnosing the abuse, fear that it may affect the reputation of their clinic, worry about what will happen to the child and his family, and unfamiliarity with child protection policy in their workplace.

The Egyptian law obligates dentists to report any suspected case of child abuse. Many studies have been published assessing dentists' knowledge and practice of CPA diagnosis and reporting. However, to our knowledge, there are no published data available about Egyptian dentists' cognition of CPA signs and diagnosis, and their actual participation in reporting suspected cases.

DETAILED DESCRIPTION:
Infants and young children are easy targets for abuse. Their challenging behaviour, defencelessness, physical weakness, and inability to escape from angry parent. They are also very young, and may not even know how to describe the injury cause. This adds additional burden to the dentist to diagnose and report such cases.

The damage that will inflict upon the child whether it is developmental, physical or mental will depend mainly on the child's age, and the scope of the abuse. The intervention to protect children isn't the responsibility of a single institute or profession, it's a shared community duty.

Risk factors for child to be subjected to abuse depend mainly on age and sex. Younger children are at greater risk for physical abuse, while older children who reached adolescence are subjected more to sexual abuse. Boys are victims of beating or physical punishment, while girls are subjected to infanticide, sexual abuse, educational and nutritional neglect. Other risk factors include poverty, being raised by single parent or very young parents, and presence of other violent relationship at home.

Studies have shown that orofacial injuries are common in case of physical abuse. From fifty to seventy-seven percent of abused children had suffered from orofacial injuries. This high percent to the head, face, and neck regions enhances the theory that easy accessibility and psychological importance of these area make them frequent target to the abuser.

Orofacial injuries due to physical abuse may include bruising, contusion, abrasions or laceration to soft tissue, dental fractures and dislocation, dental avulsion, maxillary and mandibular fractures. Skin injuries include ecchymosis and excoriations, which are commonly associated with abrasions, contusions or lacerations. These injures may be produced by natural ways like fists or slaps, instruments like household utensils, and ligature instruments like belts and shoelace.

Since orofacial injuries is common in case of CPA, and dentists are the first to examine this area, they are in better place to diagnose and report such cases. In addition to that, children who are subjected to abuse or neglect have higher incidence of caries and other oral diseases.

A study compared oral health between three groups: Children who witnessed violence or are victims of abuse, children with eating disorders, and control group, found that incidence of caries and periodontal diseases are higher in children in the abuse group than the other two groups.

Abusive parents avoid going to the same paediatrician in order not to be detected, but they feel that dentists represent less threat to them. And as dentists are in perfect position to diagnose and report CPA, their knowledge and attitude toward reporting are essential factors to fulfil their legal and ethical obligation.

Unfortunately, large portion of CPA cases are undocumented and unreported. This in addition to, high prevalence of CPA, and deficient statistics that only rely on police and social workers reports, has changed some countries policies. In America, any close contact to the child like teachers and health care workers must report suspected cases. In Europe even normal citizen can report such cases.

In a recent study navigating experience of dental professionals in UK, there was a remarkable gap between diagnosing CPA and reporting it. While 67% suspected abuse during their career, only 29% made a child protection referral. The under-reporting of CPA is also an international issue.

Although failing to diagnose cases of child physical abuse may lead to catastrophic events, dentists should be trained to know benign conditions that may be mistaken for child abuse; so that unnecessary distress is avoided. It was found that dentists who joined professional training problem can differentiate between cases of abuse and accidental injury, they were also better at discussing this sensitive topic with the parents.

The result of this study will enhance the importance of adding child abuse diagnosis and reporting methods, physical and behavioural indicators of child abuse, as well as techniques of history taking and documentation of suspected cases to pregraduate and postgraduate curriculums, increasing the dentists' awareness about their legal and ethical obligation to report suspected abuse cases. It will also help in identifying barriers to reporting CPA, and assessing dentists' training needs to make the dentists actively involved in child protection.

ELIGIBILITY:
Inclusion Criteria:

* Staff members at all departments in Faculty of Dentistry, Cairo University.
* Master's and PhD candidates enrolled at different specialities.

Exclusion Criteria:

* Intern dentists.
* Dentists who don't have a work permission in Egypt.
* Dentists who will refuse to participate.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Cluster sample, involving dentists with different experience, knowledge, age group, and specialities.
Sampling Method: Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Assessing Egyptian dentists' knowledge about child abuse diagnosis. | One month.
  Questions about the ability of dentist to diagnose abuse, using trichotomous scale (Yes/No/Don't know)
Assessing Egyptian dentists' knowledge about child abuse reporting. | One month.
  Questioning if the dentist is able to report a suspected case of child abuse, using trichotomous scale (Yes/No/Don't know)
Assessing Egyptian dentists' attitude and practice towards child abuse. | One month
  Assessment of Egyptian dentists' attitude towards child abuse reporting, and practice of reporting, using trichotomous scale (Yes/No/Don't know)

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Dabaan R, Newton JT, Asimakopoulou K. Knowledge, attitudes, and experience of dentists living in Saudi Arabia toward child abuse and neglect. Saudi Dent J. 2014 Jul;26(3):79-87. doi: 10.1016/j.sdentj.2014.03.008. Epub 2014 May 9. PMID 25057227
- [Background] Costacurta M, Benavoli D, Arcudi G, Docimo R. Oral and dental signs of child abuse and neglect. Oral Implantol (Rome). 2016 Jul 25;8(2-3):68-73. doi: 10.11138/orl/2015.8.2.068. eCollection 2015 Apr-Sep. PMID 27555907
- [Background] Harris JC, Elcock C, Sidebotham PD, Welbury RR. Safeguarding children in dentistry: 1. Child protection training, experience and practice of dental professionals with an interest in paediatric dentistry. Br Dent J. 2009 Apr 25;206(8):409-14. doi: 10.1038/sj.bdj.2009.307. PMID 19396200
- [Background] Owais AI, Qudeimat MA, Qodceih S. Dentists' involvement in identification and reporting of child physical abuse: Jordan as a case study. Int J Paediatr Dent. 2009 Jul;19(4):291-6. doi: 10.1111/j.1365-263X.2009.00971.x. Epub 2009 May 20. PMID 19476516
- [Background] Cairns AM, Mok JY, Welbury RR. Injuries to the head, face, mouth and neck in physically abused children in a community setting. Int J Paediatr Dent. 2005 Sep;15(5):310-8. doi: 10.1111/j.1365-263X.2005.00661.x. PMID 16128994
- [Background] Jordan A, Welbury RR, Tiljak MK, Cukovic-Bagic I. Croatian dental students' educational experiences and knowledge in regard to child abuse and neglect. J Dent Educ. 2012 Nov;76(11):1512-9. PMID 23144487
- [Background] Kirankumar SV, Noorani H, Shivprakash PK, Sinha S. Medical professional perception, attitude, knowledge, and experience about child abuse and neglect in Bagalkot district of north Karnataka: a survey report. J Indian Soc Pedod Prev Dent. 2011 Jul-Sep;29(3):193-7. doi: 10.4103/0970-4388.85807. PMID 21985873
- [Background] Laud A, Gizani S, Maragkou S, Welbury R, Papagiannoulis L. Child protection training, experience, and personal views of dentists in the prefecture of Attica, Greece. Int J Paediatr Dent. 2013 Jan;23(1):64-71. doi: 10.1111/j.1365-263X.2012.01225.x. Epub 2012 Mar 16. PMID 22429739
- [Background] Mogaddam M, Kamal I, Merdad L, Alamoudi N. Knowledge, attitudes, and behaviors of dentists regarding child physical abuse in Jeddah, Saudi Arabia. Child Abuse Negl. 2016 Apr;54:43-56. doi: 10.1016/j.chiabu.2016.02.004. Epub 2016 Mar 15. PMID 26990176
- [Background] Sonbol HN, Abu-Ghazaleh S, Rajab LD, Baqain ZH, Saman R, Al-Bitar ZB. Knowledge, educational experiences and attitudes towards child abuse amongst Jordanian dentists. Eur J Dent Educ. 2012 Feb;16(1):e158-65. doi: 10.1111/j.1600-0579.2011.00691.x. Epub 2011 May 5. PMID 22251340
- [Background] Ellis C. Summary of: the Scottish dental practitioner's role in managing child abuse and neglect. Br Dent J. 2013 May;214(9):454-5. doi: 10.1038/sj.bdj.2013.461. No abstract available. PMID 23660905
- [Background] Harris CM, Welbury R, Cairns AM. The Scottish dental practitioner's role in managing child abuse and neglect. Br Dent J. 2013 May;214(9):E24. doi: 10.1038/sj.bdj.2013.435. PMID 23660928